CLINICAL TRIAL: NCT06369779
Title: Clinical Evaluation of Class I and II Cavities Restored With the Combination of a New Flowable and a New Sculptable Universal Bulk-fill Composite: A Prospective Single Arm Study
Brief Title: Clinical Evaluation of a New Flowable and a New Sculptable Universal Bulk-fill Composite for Direct Restorative Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTCS 36406866
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-07

CONDITIONS: Insufficient Dental Filling or Primary Caries (Class I or II Cavities in Premolars or Molars)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (TM Fill in combination with TM Flow) (Experimental): TM Fill an TM Flow are used for restoration of class I and class II cavities
  Interventions: Device: TM Fill in combination with TM Flow

INTERVENTIONS:
Device: TM Fill in combination with TM Flow — The newly developed resin composites (TM Flow in combination with TM Fill) will be used for the restoration of class I and II cavities (3 seconds light-curing mode, 3000 milliwatt per square centimeter).

SUMMARY:
The overall objective of this clinical investigation is to evaluate the clinical safety and performance of the new flowable composite TM Flow and the new sculptable composite TM Fill for restoration of class I and class II cavities. The fillings are assessed according to selected FDI (Fédération Dentaire Internationale) criteria at baseline (7-10 days after placement of filling) and after 1, 6, 12, 24, 36 and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Age: 18-65 years
* Indication Class I or II direct restorations in premolars or molars (Replacement of insufficient fillings due to secondary caries, fractures, insufficient marginal adaptation, loss of filling or primary caries)
* Cavity width must be at least half of the cusp tip distance
* Vital teeth, regular sensitivity
* Sufficient language skills
* No active periodontits
* Preoperative VAS (visual analogue scale) values < 3 regarding tooth sensitivity and biting

Exclusion Criteria:

* Sufficient isolation of the cavity not possible
* Not completed hygiene phase or poor oral hygiene
* Missing antagonist, non-occlusion
* Missing tooth adjacent to the tooth to be treated
* Restorations replacing more than 1 cusp
* Caries profunda or very deep cavity
* Patients with a proven allergy to ingredients of the used materials (methacrylates) or local anesthetics (Articain, sulfite)
* Patients with severe systemic diseases
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ivoclar Vivadent AG, Schaan, Liechtenstein, Liechtenstein

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Restorations
Period: Overall Study
Arm/Group | Test group (TM Fill in combination with TM Flow)
Started | 65; 65 Restorations
Completed | 64; 64 Restorations
Not Completed | 1; 1 Restorations

BASELINE CHARACTERISTICS:
Arm/Group | Test group (TM Fill in combination with TM Flow)
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Hypersensitivity
Description: assessed by tests with thermal stimuli and occlusal forces (during biting) determined by VAS (Visual Analog Scale, 0 "No pain at all" - 10 "The worst pain imaginable") following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable" FDI 1: no complaint FDI 2: minor complaint FDI 3: distinct pain FDI 4: persistent pain for prolonged period of time FDI 5: treatment unavoidable
Time Frame: 1 month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Test group (TM Fill in combination with TM Flow)
Number analyzed (Participants) | 64
Number analyzed (Restorations) | 64
Restorations
  FDI Score 1 | 63
  FDI Score 2 | 0
  FDI Score 3 | 1
  FDI Score 4-5 | 0

2. Secondary Outcome: Evaluation of Functional (e.g. Fracture of the Material and Retention), Biological (e.g. Caries at Restoration Margins) and Aesthetic (e.g. Color Match) Properties of the Restorations
Description: will be assessed according to FDI criteria (grade 1-5)
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 Month Recall
Arm/Group | Test group (TM Fill in combination with TM Flow)
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT06369779/Prot_SAP_002.pdf